CLINICAL TRIAL: NCT06034717
Title: Mid Term&Short Term Outcomes in Pediatric Patients With Hemodialysis Access
Brief Title: Primary Patency in Pediatric Patients With Hemodialysis Access
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alaa Gameil Abd El-salam Hussien (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Alaa Gameil Abd El-salam Hussien, : Alaa Gameil Abd El-salam Hussien, Assiut University
Organization: Assiut University (Other)
Other Study IDs: observational
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: The Aim of This Study is to Follow up Short Term "3-6 Months"& Mid Term" 6-12months "Outcomes of Vascular Access" Native and Synthetic "in ESRD Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — pediatric patients with hemodialysis access
  All data will be collected from the study patients by the applicant. most data will be related to the patient's relative risk factors, duplex US,and physical examination and investigations. the operative details and data related to the post management follow up. this will be done under close supervision of my supervisors at the department of Vascular & EndovascularSurgery, Assiut University Hospitals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vascular access in the pediatric hemodialysis patients is a challenging,but necessary. It requires proper advance planning to assure that the best permanent access is placeds long life span. It is imperative to have a long-term vision to decrease morbidity in this unique patient population.

DETAILED DESCRIPTION:
Recent data indicate that the incidence of end stage renal disease (ESRD) in pediatrics has increased over the past two decades[1]. Hemodialysis continues to be the most frequently utilized modality for renal replacement therapy in pediatric ESRD patients One of the most challenging aspects of kidney replacement therapy in children is the creation and maintenance of a functioning vascular access to provide adequate blood flow for uremic solute removal during haemodialysis, whilst minimizing the risk of systemic infections and preserving vascular access choices for future dialysis. There are three common forms of vascularaccess: tunnelled cuffed lines placed in a central vein, arteriovenous fistulas and arteriovenous grafts using prosthetic or biological material. arterio-venous fistula"nativevascularaccesses" are the preferred vascularaccess for children on hemodialysis. Compared with a CVL, a functional artirio-venous fistula is associated with better dialysis adequacy,significantly lowering complication rates and access failure.However, CVLs remain the most frequently used vascular access in all paediatric age groups, despite international recommendations[1-4] pediatrics with ESRD from age (1-6years) start with peritoneal dialysis, and then from age (6-18years) start to use hemodialysis The 'ideal artrio-venous fistula ' is made distally in the non-dominant arm,e.g. a radiocephalic AVF, and suitable vessels are veins>2 mm and arteries > 1 mm [5,6]. Apart from vessel size,many other factors should be considered when deciding which access to create e.g. psychological preparation of the child/parent, surgical expertise, child size/weight, quality of veins,cosmetic concerns for the teenager and hand dominance for the child who wishes to self-cannulate. Maintaining the confidence of the child, parent and dialysis nursing team is vitalwhen forming the access.

thisisdone by the aid ofduplexultrasound to assess size of vein,sizeofartery,patencyofcentralvenoussystem physical examination to assess blood pressure it's important to maintain blood pressure >120,<160 to allow patency of vascular access.All thisisimportant tominimize/avoid the prolonged use of CVCs due to risks ofinfection and the need for vessel preservation. we need to use good clinical judgment when choosing the appropriate vascular access in each patient.

possible complications that can occur affecting patency of vascular access include:

1. Stenosis(Stenosis is a common complication which may affect the function of an AVF, it is the main cause of arterio-venousfistula thrombosis and failure) [7]

   . Factors that predispose to the formation of venous neo-intimal hyperplasia and stenoses include the Following: surgical injury, recurrent traumatic cannulaltion (leading to defective vascularre modelling), high blood flow inducing endothelial cell dysfunction andshear stress. Stenoses commonly present clinically with inadequate pump speed, poor dialysis adequacy or a prolonged post-dialysis bleeding time. Physical examination should be correlated with a Doppler ultrasound assessment to investigate any clinically significant stenosis. In the absence of any clinical issues, an arterio-venous fistula stenosis is considered significant if there is >20% reduction from baseline volume
2. arterio-venous fistula thrombosis Acute vascularaccess thrombosis accounts for 20-25% of all hospitalizations for hemodialysis patients and this leads to considerable morbidity and cost to healthcare providers. [8, 9] An important consideration in preventing early thrombosis peri-arterio-venousfistula formation is to maintain adequate intravascular voume. This can be achieved by reducing the ultrafiltration for a few haemodialysis sessions just after arterio-venous fistula creation and allowing permissive hypertension. Adjusting anti hypertensive treatment in this early post-operative period to maintainbloodpressure(>130). D-dimers may help guide anti-thrombotic therapy and prevent clotting.In a paediatric study, the levels of D-dimers were inversely correlated with patency rates -based protocol to prevent early arterio-venous fistula failure compared with historical controls and showed a lower rate of early thrombosis .
3. Infections Infection rates for native and synthetic vascularaccess are substantially lower (up to 10 times) than those for CVLs.. Importantly, 80% of the vascular accesses remained functional after treating the infection[10].

Haemodynamic issues High-output cardiac failure is occasionally seen in adults but is uncommon in children and is managed with arterio-venous fistula volume flow reduction . Steal syndrome ] occurs when a significant proportion of cardiac output is diverted from the distalcapillary bed by the proximal arterio-venous fistula, causing distal ischemia [11,12]. This is also rare but may require surgical revision to preserve the access and alleviate the distal ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* ) Ages :6-18 2) gender: All 3) Children on regular dialysis 4)children with duplex criteria including: vein >2mm artery>1mm patent , respirophasic central venous system 5) children's parents compliance to follow-up.

Exclusion Criteria:

1)Children with ESRD contraindicated for vascular intervention including: Children with resistance hyper-tention Children with medical history of bleeding tendency Children with hyper-coagulable state 2)children with duplex criteria including: vein fibrotic "<2mm" artery<1mm occluded central veins 3)Children's parents not compliance to follow up

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients fulfilling the inclusion and exclusion criteria will be included in this study with time frame 1year
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-09-28 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to follow up Short term "3-6 months"& Mid term" 6-12months "outcomes of Vascular access" native and synthetic "in ESRD pediatrics | from 1october 2022to 28september 2023
  evaluation of short term "3-6months" and Mid term "6-12months" outcomes, patterns of complication in pediatrics with hemodialysis access(time frame one year after surgey) Primary (unassisted) patency The interval from the time of access creation until the first access thrombosis or any intervention to maintain or restore blood flow

SECONDARY OUTCOMES:
2ry patency | from 1october 2022to 28september 2023
  To identify possible complications&how to avoid Secondary (cumulative) patency "The time from access creation until access abandonment".
  Functional secondary patency" The interval from the first successful two-needle cannulation for haemodialysis treatment to access abandonment" possible complications include:
  1. Stenosis
  2. thrombosis
  3. Infections

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university hospital, Asyut, Egypt